CLINICAL TRIAL: NCT00477412
Title: Phase I/II Study of Bortezomib (VELCADE) Plus Rituximab-HyperCVAD Alternating With Bortezomib Plus Rituximab-High Dose Methotrexate/Cytarabine in Patients With Untreated Aggressive Mantle Cell Lymphoma
Brief Title: Bortezomib, Rituximab and Combination Chemotherapy in Treating Participants With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0697; NCI-2018-01851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0697 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Methotrexate; merphos; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Participants receive Drug Combination I during courses 1, 3, 5, and 7 (if needed) and Drug Combination II during courses 2, 4, 6, and 8 (if needed) in the absence of disease progression or unacceptable toxicity.
  Drug Combination I: Participants receive rituximab IV over 6 hours on day 1, cyclophosphamide IV over 3 hours BID on days 2-4, doxorubicin IV over 15-30 minutes on day 5, vincristine IV over 15-30 minutes on days 5 and 12, dexamethasone PO or IV on days 2-5 and 12-15, and bortezomib IV over a few seconds after the first dose of cyclophosphamide and immediately after vincristine and doxorubicin have been given on day 5.
  Drug Combination II: Participants receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours every 12 hours on days 3-4.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Methotrexate; Biological: Rituximab; Drug: Vincristine

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine — Given IV
  Other Names: LEUROCRISTINE; VCR; Vincrystine

SUMMARY:
This phase I/II trial studies the side effects and best dose of bortezomib when given with rituximab and chemotherapy drugs and to see how well they work in treating participants with mantle cell lymphoma. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, dexamethasone, methotrexate, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving bortezomib, rituximab and combination chemotherapy may work better at treating mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and the maximum tolerated dose (MTD) of bortezomib when added to the combination of rituximab, methotrexate, and cytarabine alternating with bortezomib, rituximab-hyperfractionated cyclophosphamide, vincristine, doxorubicin, dexamethasone (hyperCVAD) in patients with untreated aggressive mantle cell lymphoma. (Phase I) II. Evaluate the time to failure (TTF) rate following therapy with bortezomib plus rituximab-hyperCVAD alternating with bortezomib plus rituximab-high dose methotrexate/cytarabine in patients between 18 and 79 years of age with untreated aggressive mantle cell lymphoma. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate overall response rate, complete remission rate, overall survival, and duration of remission. (Phase I) II. Evaluate overall response rate, overall survival, and duration of remission. (Phase II) III. Evaluate toxicity of the combination regimen. (Phase II) IV. Correlate outcome with pretreatment markers. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of bortezomib followed by a phase II study.

Participants receive Drug Combination I during courses 1, 3, 5, and 7 (if needed) and Drug Combination II during courses 2, 4, 6, and 8 (if needed) in the absence of disease progression or unacceptable toxicity.

Drug Combination I: Participants receive rituximab intravenously (IV) over 6 hours on day 1, cyclophosphamide IV over 3 hours twice daily (BID) on days 2-4, doxorubicin IV over 15-30 minutes on day 5, vincristine IV over 15-30 minutes on days 5 and 12, dexamethasone orally (PO) or IV on days 2-5 and 12-15, and bortezomib IV over a few seconds after the first dose of cyclophosphamide and immediately after vincristine and doxorubicin have been given on day 5.

Drug Combination II: Participants receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours every 12 hours on days 3-4.

After completion of study treatment, participants are followed up every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of previously untreated nodular or diffuse mantle cell lymphoma and their blastoid cytologic variant.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Serum bilirubin < 1.5 mg/dl and serum creatinine < 2.0 mg/dl within 14 days before enrollment (unless higher levels are due to lymphoma).
* Platelet count > 100,000/mm^3 within 14 days before enrollment (unless due to lymphoma).
* Absolute neutrophil count (ANC) > 1,000/mm^3 within 14 days before enrollment (unless due to lymphoma).
* Cardiac ejection fraction >= 50% by echocardiogram (ECHO) or multigated acquisition (MUGA).
* Patients must be willing to receive transfusions of blood products.
* Voluntary written Institutional Review Board (IRB)-approved informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal for at least 1 year before the Screening visit or surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of birth control, at the same time (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from the time of signing the informed consent through 30 days after the last dose of study treatment, or agree to completely abstain from heterosexual intercourse.
* Male subject, even if surgically sterilized (ie, status post vasectomy) agrees to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study treatment, or agree to completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Human immunodeficiency virus (HIV) infection.
* Central nervous system (CNS) involvement.
* Co-morbid medical or psychiatric illnesses that preclude treatment with intense dose chemotherapy.
* Concurrent or previous malignancy with < 90% probability of survival at 5 years.
* Patient has >= grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiography (ECG) abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Participating in clinical trials with other investigational agents not included in this trial within 14 days of the start of this trial and throughout the duration of this trial.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-04-03 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with newly diagnosed MCL were enrolled into a phase 2 trial approved by the institutional review boards of both. The University of Texas MD Anderson Cancer Center and John Theurer Cancer Center at Hackensack University.
Groups:
- Phase I Bortezomib 0.7 mg/m^2; Phase I Bortezomib 1.0 mg/m^2; Phase 1 Maximum Tolerated Dose (MTD) 1.3 mg/m^2; Phase II- Treatment (Combination Chemotherapy) 1.3 mg/m^2: Participants receive Drug Combination I during courses 1, 3, 5, and 7 (if needed) and Drug Combination II during courses 2, 4, 6, and 8 (if needed) in the absence of disease progression or unacceptable toxicity.
  Drug Combination I: Participants receive rituximab IV over 6 hours on day 1, cyclophosphamide IV over 3 hours BID on days 2-4, doxorubicin IV over 15-30 minutes on day 5, vincristine IV over 15-30 minutes on days 5 and 12, dexamethasone PO or IV on days 2-5 and 12-15, and bortezomib IV over a few seconds after the first dose of cyclophosphamide and immediately after vincristine and doxorubicin have been given on day 5.
  Drug Combination II: Participants receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours every 12 hours on days 3-4.
Period: Overall Study
Arm/Group | Phase I Bortezomib 0.7 mg/m^2 | Phase I Bortezomib 1.0 mg/m^2 | Phase 1 Maximum Tolerated Dose (MTD) 1.3 mg/m^2 | Phase II- Treatment (Combination Chemotherapy) 1.3 mg/m^2
Started | 4 | 3 | 5 | 95
Completed | 3 | 3 | 4 | 87
Not Completed | 1 | 0 | 1 | 8
Not completed — Death | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Second Malignancy | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II- Treatment (Combination Chemotherapy): Participants receive Drug Combination I during courses 1, 3, 5, and 7 (if needed) and Drug Combination II during courses 2, 4, 6, and 8 (if needed) in the absence of disease progression or unacceptable toxicity.
  Drug Combination I: Participants receive rituximab IV over 6 hours on day 1, cyclophosphamide IV over 3 hours BID on days 2-4, doxorubicin IV over 15-30 minutes on day 5, vincristine IV over 15-30 minutes on days 5 and 12, dexamethasone PO or IV on days 2-5 and 12-15, and bortezomib IV over a few seconds after the first dose of cyclophosphamide and immediately after vincristine and doxorubicin have been given on day 5.
  Drug Combination II: Participants receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours every 12 hours on days 3-4.
- Total: Total of all reporting groups
Arm/Group | Phase I Bortezomib 0.7 mg/m^2 | Phase I Bortezomib 1.0 mg/m^2 | Phase 1 Maximum Tolerated Dose (MTD) 1.3 mg/m^2 | Phase II- Treatment (Combination Chemotherapy) | Total
Number analyzed (Participants) | 4 | 3 | 5 | 95 | 107
Age, Continuous [Median (Full Range); unit: years] | 40 [18 to 65] | 40 [18 to 65] | 40 [18 to 65] | 61 [38 to 75] | 51 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 28 | 28
  Male | 4 | 3 | 5 | 67 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 13 | 13
  Not Hispanic or Latino | 4 | 3 | 5 | 55 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 27 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 4 | 3 | 5 | 66 | 78
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 27 | 27
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 5 | 95 | 107

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Bortezomib (Phase I)
Description: Determine the safety and the maximum tolerated dose (MTD) of bortezomib when added to the combination of rituximab, methotrexate, and cytarabine alternating with bortezomib, rituximab-hyperCVAD in patients with untreated aggressive mantle cell lymphoma.
Time Frame: Cycle 1 Day 1 - End of Cycle 2 up to 60 days.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1 Maximum Tolerated Dose (MTD): Participants receive Drug Combination I during courses 1, 3, 5, and 7 (if needed) and Drug Combination II during courses 2, 4, 6, and 8 (if needed) in the absence of disease progression or unacceptable toxicity.
  Drug Combination I: Participants receive rituximab IV over 6 hours on day 1, cyclophosphamide IV over 3 hours BID on days 2-4, doxorubicin IV over 15-30 minutes on day 5, vincristine IV over 15-30 minutes on days 5 and 12, dexamethasone PO or IV on days 2-5 and 12-15, and bortezomib IV over a few seconds after the first dose of cyclophosphamide and immediately after vincristine and doxorubicin have been given on day 5.
  Drug Combination II: Participants receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours every 12 hours on days 3-4.
Arm/Group | Phase 1 Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12
mg/m^2 | 1.3

2. Primary Outcome: Time to Failure (Phase II)
Description: Failure will be defined as recurrence/progression of disease or death from either disease or toxicity. Bayesian toxicity monitoring schema will be used to monitor severe toxicity profile in combined therapy. Severe toxicity is defined as at least two episodes of neutropenic fever during treatment courses.
Time Frame: First date of diagnosis up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Phase II- Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 95
months | 55 [0 to 60]

3. Secondary Outcome: Number of Participants With Overall Response Rate
Description: Response rate is determined by CT scans of the chest, abdomen, and pelvis, unilateral BM biopsy and aspirate with lymphoma markers (if initially positive) and colonoscopy/endoscopy if applicable.
Time Frame: Up to 5 years
Population: Overall Response Rate was measured in Phase II only. No data collected for Phase I.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II- Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 94
Participants | 87

4. Secondary Outcome: Overall Survival
Description: Overall survival is the time in number of months from start of study treatment to date of death due to any cause.
Time Frame: Date of diagnosis to last known date of survival, up to 5 years
Population: Overall Response Rate was measured in Phase II only. No data collected for Phase I.
Measure: Median (Full Range); unit: months
Arm/Group | Phase II- Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 94
months | 44 [1 to 60]

ADVERSE EVENTS:
Time Frame: up to 5 years
Groups:
- Phase 1 Maximum Tolerated Dose (MTD) Bortezomib 1.3 mg/m^2; Phase II- Treatment (Combination Chemotherapy): Participants receive Drug Combination I during courses 1, 3, 5, and 7 (if needed) and Drug Combination II during courses 2, 4, 6, and 8 (if needed) in the absence of disease progression or unacceptable toxicity.
  Drug Combination I: Participants receive rituximab IV over 6 hours on day 1, cyclophosphamide IV over 3 hours BID on days 2-4, doxorubicin IV over 15-30 minutes on day 5, vincristine IV over 15-30 minutes on days 5 and 12, dexamethasone PO or IV on days 2-5 and 12-15, and bortezomib IV over a few seconds after the first dose of cyclophosphamide and immediately after vincristine and doxorubicin have been given on day 5.
  Drug Combination II: Participants receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours every 12 hours on days 3-4.
Arm/Group | Phase I Bortezomib 0.7 mg/m^2 | Phase I Bortezomib 1.0 mg/m^2 | Phase 1 Maximum Tolerated Dose (MTD) Bortezomib 1.3 mg/m^2 | Phase II- Treatment (Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 4/4 | 2/3 | 5/5 | 7/94
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 1/5 | 45/94
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/5 | 94/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Bortezomib 0.7 mg/m^2 (N=4) | Phase I Bortezomib 1.0 mg/m^2 (N=3) | Phase 1 Maximum Tolerated Dose (MTD) Bortezomib 1.3 mg/m^2 (N=5) | Phase II- Treatment (Combination Chemotherapy) (N=94)
Neutropenic Fever (Infections and infestations) | 1 | 1 | 1 | 45
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Bortezomib 0.7 mg/m^2 (N=4) | Phase I Bortezomib 1.0 mg/m^2 (N=3) | Phase 1 Maximum Tolerated Dose (MTD) Bortezomib 1.3 mg/m^2 (N=5) | Phase II- Treatment (Combination Chemotherapy) (N=94)
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 4 | 94
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3 | 4 | 94
Infection (Infections and infestations) | 0 | 0 | 0 | 11
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 4
Line Infection (Infections and infestations) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 3
Mucositis (Gastrointestinal disorders) | 0 | 0 | 0 (0) | 3
Atrial Fibrillation/ Flutter (Cardiac disorders) | 0 | 1 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Sinus Infection (Infections and infestations) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Leukocytosis (Investigations) | 0 | 1 | 0 | 0
Anemia (Investigations) | 4 | 3 | 4 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Petechiae (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Leukopenia (Investigations) | 3 | 3 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Fever (Non-NP) (General disorders) | 0 | 1 | 0 | 0
Elevated ALT (Investigations) | 0 | 1 | 1 | 0
Elevated AST (Investigations) | 1 | 1 | 0 | 0
Edema (HN) (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT00477412/Prot_SAP_000.pdf